CLINICAL TRIAL: NCT05666401
Title: Does Follicle Diameter and Total Duration Spent for Oocyte Pick up Has Any Effect on Embryological Parameters and Clinical Pregnancy Rates
Brief Title: Effect of Duration and Follicle Diameter During Oocyte Pick up on Embryological Parameters
Status: Completed | Type: Observational
Sponsor: Eurofertil IVF Health Center (Other)
Responsible Party: Principal Investigator, Elif Güler Ergin, Main investigator, Eurofertil IVF Health Center
Other Study IDs: Eurofertil-OPU
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Follicle Size; Embryologic Parameters; Duration
Keywords: follicle; dimension; IVF; embryological parameters; duration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: follicles with a diameter of 17 mm and more
  Interventions: Procedure: follicle diameter and duration of procedure
- group 2: follicles with a diameter of 14 mm to 17 mm
  Interventions: Procedure: follicle diameter and duration of procedure

INTERVENTIONS:
Procedure: follicle diameter and duration of procedure — to investigate if smaller follicles thrive embryos as the bigger follicles
  Other Names: success rates

SUMMARY:
Investigators aim to investigate if the time spent for smaller follicles worth to deal with. The difference between follicle groups are recorded for embryological parameters. Results will be analysed for yielding transfer embryo and pregnancy rates between groups.

DETAILED DESCRIPTION:
There are papers about follicle dimensions and volumes studying their effect on embryologic parameters. But most of these studies are far from practical approach and are not easily applicable, such as 3D volumetric measurement is not feasible for most of the clinics. Also one of the points important for us it to evaluate the duration of the procedure and the possible positive effect of shortening the duration for better results. Investigators plan to measure the follicles just before puncture and arrange two groups. Group 1,follicles with diameter of 17 mm and more, and group 2 follicles between14-17 mm. Maturation, fertilization, cleavage characteristics are recorded. The source of chosen transfer embryo and crio-preserved embryos per cycle is also point of interest.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 year old women

Exclusion Criteria:

* History of recurrent implantation failure (RIF)
* Known chromosomal abnormality
* Severe male factor and azospermia

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — infertile women attending for IVF
Study Population: Couples attending to our clinic for IVF - ICSI without history of RIF and severe male factor
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2022-03-19 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
transfer embryo | 5 to 7 days
  comparing groups as the source of transfer embryo

SECONDARY OUTCOMES:
clinical pregnancy | 3 weeks
  comparing groups as the source of implanted embryo

CONTACTS AND LOCATIONS:
Overall Officials: gercek aydin, Study Director — bursa Eurofertil IVF center
Locations (2):
- Turkey (Türkiye) (2):
  - Bursa Eurofertil IVF center, Bursa
  - Eurofertil IVF center, Bursa

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided yet but probably be available upon request